CLINICAL TRIAL: NCT01237756
Title: Electrical Impedance Tomography for Endotracheal Tube Placement in Pediatric Patients
Brief Title: Electrical Impedance Tomography for Endotracheal Tube Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Dr. med. Daniel Steinmann, University Medical Center Freiburg
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 198/08
Record Dates: First submitted 2010-01-25; First posted 2010-11-10 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2008-06

CONDITIONS: Endotracheal Tube Placement
Keywords: pediatric anesthesia; endotracheal tube; electrical impedance tomography; misplacement; endobronchial

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- pediatric (Experimental)
  Interventions: Device: measurement of left and right lung ventilation

INTERVENTIONS:
Device: measurement of left and right lung ventilation — Patients are ventilated after endotracheal tube placement and left and right lung ventilation if determined using electrical impedance tomography
  Other Names: EIT, Draeger

SUMMARY:
Endobronchial tube misplacement is serious complication during general anesthesia in pediatric patients. Correct placement of the endotracheal tube (ETT) in the trachea is crucial. Several methods have been suggested for determination of correct ETT placement. However, to date, auscultation of the left and right lung is the standard of care and the only ubiquitary available method with an error rate of up to 12%. Electrical impedance tomography (EIT) is a new non-invasive method for evaluation of left and right lung ventilation. In this study the investigators investigate the potential role of EIT for proper placement of pediatric endotracheal tubes.

DETAILED DESCRIPTION:
Several methods have been suggested for determination of correct ETT placement. These include for example the marker method, the mainstem method or the formula method. However, to date, auscultation of the left and right lung is the standard of care and the only ubiquitary available method with an error rate of up to 12%. Electrical impedance tomography (EIT) is a new non-invasive method for evaluation of left and right lung ventilation. In this study the investigators investigate the potential role of EIT for proper placement of pediatric endotracheal tubes. For this purpose, pediatric patients are routinely intubated for cardiac catheterization using the mainstem method or 3xETT size method. Placement of the ETT is then verified by intraoperative fluoroscopy and lung ventilation is verified by EIT.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent from the parents
* endotracheal intubation with a standard endotracheal tube

Exclusion Criteria:

* refusal of written informed consent
* severe lung diseases
* contraindication for use of electrical impedance tomography

Ages: 1 Week to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2008-09; Primary Completion 2009-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
determination of proper endotracheal tube placement | endotracheal tube placement is immediately verified after endotracheal intubation with fluoroscopy and electrical impedance tomography during the general anesthesia for cardiac catheterization

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Steinmann, MD, Principal Investigator — University Medical Center Freiburg
Locations (1):
- University Medical Center Freiburg, Freiburg im Breisgau, Germany

REFERENCES:
- [Background] Steinmann D, Stahl CA, Minner J, Schumann S, Loop T, Kirschbaum A, Priebe HJ, Guttmann J. Electrical impedance tomography to confirm correct placement of double-lumen tube: a feasibility study. Br J Anaesth. 2008 Sep;101(3):411-8. doi: 10.1093/bja/aen166. Epub 2008 Jun 17. PMID 18559350